CLINICAL TRIAL: NCT05623774
Title: A Dose Calibration and Dose Equivalence Pharmacokinetic Study in Healthy Volunteers Comparing IkT-001Pro to Imatinib Mesylate 400mg
Brief Title: A Dose Calibration Study Comparing IkT-001Pro to Imatinib Mesylate 400mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inhibikase Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IkT-001Pro-501
Record Dates: First submitted 2022-11-09; First posted 2022-11-21 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: CML
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Intervention Model Description: This is a crossover design dose calibration study in healthy volunteers to identify a dose of IkT-001Pro film-coated tablets that would be equivalent to imatinib free base 400 mg film-coated tablets containing imatinib mesylate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Calibration (Active Comparator): In Part A, cohorts will consist of 8 subjects who will receive a single dose of Ikt-001Pro and then cross over to a single does of imatinib following a 7 day washout.
  Interventions: Drug: Imatinib Mesylate; Drug: IkT-001Pro
- Dose Equivalance (Active Comparator): In Part B, up to 16 subjects will receive IkT001-Pro and up to 16 subjects will receive 400mg of imatinib mesylate. After a 7 day washout period the subjects will switch to receive the drug they did not previously receive.
  Interventions: Drug: Imatinib Mesylate; Drug: IkT-001Pro
- Dose Equivalence at 600 mg): (Active Comparator): In Part C, up to eight (8) subjects will be administered a single dose of 800 mg IkT-001Pro. After a 7-day washout period, the subjects will switch to 600 mg imatinib.
  Interventions: Drug: Imatinib Mesylate; Drug: IkT-001Pro

INTERVENTIONS:
Drug: Imatinib Mesylate — 400mg tablet
Drug: IkT-001Pro — 100mg or 400mg tablet

SUMMARY:
This study investigates the safety, tolerability and dose equivalence of drug IkT-001Pro in healthy volunteers (18 to 55 years old) in comparison to imatinib mesylate. This study is designed in 3 parts.

Part A consists of 3 cohorts. In cohort 1 healthy participants will take a single, oral dose of 400mg IkT-001Pro then will be followed by a single dose of 400mg Imatinib mesylate after a 7-day washout. Cohort 2 and 3 will follow the same structure as cohort 1 with a different Ikt-001Pro dose.

Part B will be chosen using Part A data by statistical procedures. Part B will enroll 32 subjects to demonstrate the bioequivalence of IkT-001Pro (the 'Test') to 400 mg imatinib delivered as imatinib mesylase (the 'Reference').

Part C (Dose Equivalence at 600 mg):

Part C will enroll up to eight (8) subjects to demonstrate bioequivalence of imatinib delivered as 800 mg IkT-001Pro (the 'Test') to 600 mg imatinib delivered as imatinib mesylate ('the Reference')

DETAILED DESCRIPTION:
Part A, Dose Calibration Cohort:

This is a crossover design dose calibration study in healthy volunteers to identify a dose of IkT-001Pro film-coated tablets that would be equivalent to imatinib free base 400 mg film-coated tablets containing imatinib mesylate.

Dose calibration cohorts will each consist of eight (8) subjects who will receive a single dose of IkT-001Pro at 400, 500 or 600 mg and then crossover to a single dose of imatinib 400 mg delivered as imatinib mesylate following a 7-day washout. The three cohorts will have staggered starting points. The 400 mg IkT-001Pro dose, washout and 400 mg imatinib delivered as imatinib mesylate will be completed first including full PK analysis. Following review of the PK data at 400 mg IkT-001Pro, the 500 mg and 600 mg cohorts will be enrolled approximately simultaneously.

Pharmacokinetic plasma samples for all three cohorts will be drawn pre-dose at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours after dosing. A 7-day washout period will take place between dosing of IkT-001Pro and dosing of 400 mg imatinib delivered as imatinib mesylate. PK plasma samples for the imatinib mesylate arm will be obtained on the same sampling schedule as the IkT-001Pro arm.

Part B- Dose Equivalence Cohort:

Part B will test the bioequivalence of the IkT-001Pro dose chosen in Part A. In this two-period crossover design dose equivalence study, up to 16 subjects will receive IkT-001Pro and up to 16 subjects will receive 400 mg imatinib as imatinib mesylate as a single dose. The dose of IkT-001Pro will be computed from the exposures measured in Part A to estimate the dose of IkT-001Pro that should be equivalent to 400 mg imatinib delivered as imatinib mesylate. After a 7-day washout period, the subjects that began on IkT-001Pro will switch to 400 mg imatinib delivered as imatinib mesylate. Similarly, the subjects that began on 400 mg imatinib delivered as imatinib mesylate will switch to the equivalent dose of IkT-001Pro. Blood samples for PK assessment will be drawn pre-dose and 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hours after dosing for both IkT-001Pro and 400 mg imatinib.

Part C- Dose Equivalence at 600 mg:

Part C will test the single dose bioequivalence of imatinib free base delivered as the equivalent dose IkT-001Pro dose computed from Part A to single dose of imatinib delivered as 600 mg imatinib mesylate. Up to eight (8) subjects will be administered a single dose of 800 mg IkT-001Pro. After a 7-day washout period, the subjects will switch to 600 mg imatinib free base delivered as imatinib mesylate.

Blood samples for PK assessment will be drawn pre-dose and 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16, 24, 48, 72 and 96 hrs post-dose on Day 1. The same sampling schedule will be followed for the IkT-001Pro and imatinib mesylate dosing periods.

General Methodological Considerations:

The Dose Calibration and Dose Equivalence cohorts will consist of up to 14 visits over a period of up to 28 days prior to dosing and 28 days after dosing. The dose-escalation pattern and timing for IkT-001Pro in Part A or Part B may be modified by the Safety Review Committee (SRC).

Subjects in each cohort of the study will be admitted to the unit approximately 24 hours prior to the expected time of dosing. They will be confined to the unit for approximately 96 hours in Part A and Part B of the study for each drug product to be administered. Subjects will not be confined to the unit during the wash-out period. No subject may be discharged from the unit until the investigator is satisfied that they have no continuing adverse events that could be related to study drug.

A full breakfast must be given no more than 60 mins prior to dosing in Parts A and B. The meal must be a high-fat (approximately 50 percent of total caloric content of the meal) and high-calorie (approximately 800 to 1000 calories) meal. The meal should derive approximately 150, 250, and 500-600 calories from protein, carbohydrate, and fat, respectively. The caloric breakdown of the meal must be provided in the study report. The single dose of IkT-001Pro or 400 imatinib delivered as imatinib mesylate is to be taken after the meal with a large glass of water (240 ml or 8 oz).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have all questions about the study answered and must have signed the informed consent document before any study-specific procedures are performed.
2. Healthy ambulatory male and female subjects > 18 to < 55 years of age at the Screening visit, with no history or evidence of clinically relevant medical disorders as determined by the Investigator in consultation with the Sponsor.
3. Bodyweight > 50 kg and body mass index (BMI) > 18.0 and < 32.0 kg/m2 at the screening visit.
4. Physical examination, clinical laboratory values, vital signs, and electrocardiogram (ECG) data. Vital signs and clinical laboratory values must be within the normal range and or deemed not clinically significant by the PI and ECG tracings must be normal at baseline and/or deemed not clinically significant by the PI.
5. Female subjects must be postmenopausal, permanently sterile (bilateral tubal occlusion), or of childbearing potential with a negative pregnancy test, non-breastfeeding, and using two highly effective methods of birth control prior to screening and through completion of the last follow-up visit. If a subject discontinues early after receiving a dose of study drug, she must continue this method of birth control for at least 7 days following the last dose of the study drug. Highly effective methods of birth control are defined as follows: hormonal (ie, established use of oral, implantable, injectable, or transdermal hormonal methods of contraception); placement of an intrauterine device; placement of an intrauterine system; and mechanical /barrier method of contraception (ie, condom or occlusive cap [diaphragm or cervical/vault cap] in conjunction with spermicide [foam, gel, film, cream or suppository]).
6. Male subjects must agree to practice an acceptable method of highly effective birth control from the Screening visit, while on study and for 7 days after receiving the last dose of study drug. Highly effective methods of birth control include sexual abstinence; vasectomy; or a condom with spermicide (men) in combination with their partner's highly effective method.
7. Males must be willing to abstain from sperm donation from the screening visit, while on study and through 30 days after receiving the last dose of study drug.

Exclusion Criteria:

1. Any subject with previous exposure to imatinib or known hypersensitivity to imatinib.
2. Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at the screening and admission visits. Abnormalities considered to be non-clinically significant by the Investigator are acceptable.
3. Clinically significant abnormal physical examination or 12-lead electrocardiogram (ECG) at the screening or admission visits. NOTE: QTcF interval of > 450 msec in males or > 470 msec in females will be the basis for exclusion from the study. ECG may be repeated for confirmatory purposes if initial values obtained exceed the limits specified.
4. Clinically significant abnormal renal function defined as a creatinine clearance rate < 90 mL/min
5. Significant history (within six months prior to receiving the study drug) and/or presence of hepatic, renal, cardiovascular, pulmonary, gastrointestinal, endocrinological, hematological, dermatological, psychiatric, neurological, immunologic, ophthalmologic, metabolic, fluid retention and edema, bleeding disorders including hemorrhage or oncological disease.
6. Any subject with a history, presence and/or current evidence of serologic positive result for hepatitis B surface antigen, hepatitis C antibodies, or HIV antibodies 1 or 2.
7. Recent history (within previous six months prior to screening) of alcohol or drug abuse (as judged by the investigator), or has consumed > 2 alcohol drinks/day during the last three months prior to screening (one glass is approximately equivalent to: beer [284 mL], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]). Subjects that consume three glasses of alcoholic beverages per day but less than 14 glasses per week may be enrolled at the discretion of the Investigator. Positive screens for alcohol or controlled substances at the screening or admission visits will disqualify a subject from study participation.
8. Any subject who currently uses or has regularly used tobacco or tobacco-containing products (cigarettes, pipes, etc.) for at least 30 days prior to screening or positive urine cotinine screen (>300 ng/mL) at the screening or admission visits.
9. Any subject who has received treatment with an investigational drug during the 30 days prior to screening. Exposure to an investigational medical device within 30 days of screening.
10. Use of agents known to affect drug metabolism: use of any known CYP3A4 inducers and/or inhibitors or consumed grapefruit juice, grapefruit, Seville oranges or St John's Wort or products containing these within 14 days prior to first administration of study drug. Strong inducers of CYP3A4 include dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifampicin and phenobarbital. Strong inhibitors of CYP3A4 include ketoconazole, itroconazole, clarythromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin and voriconazole.
11. Investigative site personnel or their immediate families (spouse, parent, child or sibling whether biological or legally adopted).
12. Any subject unwilling or unable to comply with study procedures.
13. Pregnant or nursing women.
14. Anyone who does not meet the requirements for exclusion of certain concomitant medications as defined in Section 7.5.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Exposure of imatinib after administration of IkT-001Pro and imatinib mesylate, as measured by area under the concentration-time curve for imatinib from time zero to last measurable concentration (AUC(0-last)) | Day 1 through day 12
  Area under the concentration-time curve for imatinib from time zero to last measurable concentration (AUC0-last)
Exposure of imatinib after administration of IkT-001Pro and imatinib mesylate, as measured by area under the concentration-time curve for imatinib from time zero to infinity (AUC0-inf) | Day 1 through day 12
  Area under the concentration-time curve for imatinib from time zero to infinity (AUC(0-inf))
Exposure of imatinib after administration of IkT-001Pro and imatinib mesylate, as measured by the maximum plasma concentration (Cmax) of imatinib | Day 1 through day 12
  The maximum plasma concentration (Cmax) of imatinib
Safety: Incidence and temporal profile of treatment-emergent adverse events (TEAEs) evaluated by type/nature, severity/intensity, seriousness, and relationship to study intervention | Day 1 through day 12
  Incidence and temporal profile of treatment-emergent adverse events (TEAEs)
Safety: Proportion of those in each dosing cohort who discontinued the assigned regimen | Day 1 through day 12
  Proportion of those in each dosing cohort who discontinued the assigned regimen

SECONDARY OUTCOMES:
Exposure of imatinib after administration of IkT-001Pro and imatinib mesylate, as measured by imatinib pharmacokinetic parameters for terminal rate constant | Day 1 through day 12
  Measurement of lamda-z
Exposure of imatinib after administration of IkT-001Pro and imatinib mesylate, as measured by imatinib pharmacokinetic parameters for terminal half-life | Day 1 through day 12
  Measurement of terminal half-life t1/2
Exposure of imatinib after administration of IkT-001Pro and imatinib mesylate, as measured by imatinib pharmacokinetic parameters for time to maximum concentration | Day 1 through day 12
  Time to reach maximum concentration (tmax)
Exposure of imatinib after administration of IkT-001Pro and imatinib mesylate, as measured by imatinib pharmacokinetic parameters for dose normalized maximum concentration | Day 1 through day 12
  Dose-normalized maximum concentration Cmax/D, where D is the dose in mg
Exposure of imatinib after administration of IkT-001Pro and imatinib mesylate, as measured by imatinib pharmacokinetic parameters for dose normalized area under the time concentration curve to last time point | Day 1 through day 12
  Dose-normalized AUC(0-t)/D, where D is the dose in mg
Exposure of imatinib after administration of IkT-001Pro and imatinib mesylate, as measured by imatinib pharmacokinetic parameters for dose-normalized area under the time concentration curve from 0 to infinite time | Day 1 through day 12
  Dose-normalized AUC(0-infinity)/D, where D is the dose in mg.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Valentine, DO, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No